CLINICAL TRIAL: NCT01976507
Title: Use of Dabigatran Etexilate to Prevent Stroke and Thromboembolism in Patients Undergoing Left Atrial Catheter Ablation Procedures for Paroxysmal or Persistent (Non-permanent) Atrial Fibrillation and Left Atrial Flutter
Brief Title: Use of Dabigatran Etexilate to Prevent Stroke and Thromboembolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Christopher Ellis, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 121204
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Results first posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dabigatran etexilate mesylate (Experimental): Immediately following the ablation procedure (4-6 hours after sheath pull and vascular hemostasis), dabigatran etexilate 150mg bid, or 75mg twice daily based on creatinine clearance in the Use in Specified Populations (USPI), will be administered for a minimum of 3 months post RF ablation.
  Interventions: Drug: dabigatran etexilate mesylate

INTERVENTIONS:
Drug: dabigatran etexilate mesylate — Immediately following the ablation procedure (4-6 hours after sheath pull and vascular hemostasis), dabigatran etexilate 150mg bid, or 75mg twice daily based on creatinine clearance in the Use in Specified Populations (USPI), will be administered for a minimum of 3 months post RF ablation.
  Other Names: Pradaxa

SUMMARY:
The purpose of this study is to evaluate major adverse bleeding risks, and thromboembolic event rates post radiofrequency (RF) ablation. The primary goal is to establish safety of dabigatran use for peri-procedural anti-coagulation after left atrial catheter radiofrequency ablation, or cryoablation procedures.

DETAILED DESCRIPTION:
Study design

Approximately 100 patients who plan to have pulmonary vein isolation by antral radiofrequency or cryoablation for paroxysmal or persistent atrial fibrillation, or left atrial flutter following prior left atrial ablation procedures, with CHADS2 score of 0-6 or CHADS2-VASc score 0-9 will be eligible for this trial and enrolled. A transesophageal echocardiogram (TEE) will be performed pre-procedure based on the presenting cardiac rhythm the day of planned catheter ablation, stroke risk by CHADS2 or CHADS2-VASc score, and preceding use of therapeutic anti-coagulation (as per current 2012 HRS/ACC/ESC guidelines on atrial fibrillation management). Immediately following the ablation procedure (4-6 hours after sheath pull and vascular hemostasis), dabigatran etexilate 150mg bid, or 75mg twice daily based on creatinine clearance in the Use in Specified Populations (USPI), will be administered for a minimum of 3 months post RF ablation. This represents the standard blanking period for post atrial fibrillation or left atrial flutter catheter ablation anticoagulation therapy. After the 3 months blanking period, patients may safely be taken off dabigatran in the low risk group for stroke or thromboembolism, according to the investigators discretion (CHADS 2 score 0-1, or CHADS2-VASc score 0-1). If on dabigatran etexilate pre-procedure, the drug will be held at least 24 hours before the intervention depending on renal function of the patient (as per recommendations in the USPI). If possible, discontinue dabigatran 1 to 2 days (CrCl >50 mL/min) or 3 to 5 days (CrCl <50 mL/min) before an invasive or surgical procedure, due to increased risk of bleeding.

Dabigatran etexilate will be resumed 4-6 hours after sheath pull and vascular hemostasis post ablation as above. Intra-procedure intravenous heparin drip will be started once left atrial access is obtained with an ACT goal target 300-350 seconds by weight based nomogram. Standardized ablation endpoints (4 vein entrance and exit block with post ablation adenosine challenge and/or isoproterenol, or termination of left atrial flutter and completion of linear ablation confirmed by differential pacing) will be documented, along with radiofrequency or cryoablation

delivery time, fluoroscopy and total case time. Inpatient adverse events will be documented, and outpatient follow up will occur at 1 and 3 months post ablation per standard protocol, with documentation of all composite endpoints (see below). In addition, a 30 day post study phone call follow up will be performed (30 days +/- 4 days following the 3 month visit). Please see Table 1 for the schedule of events.

Our hypothesis is that exposure to dabigatran in the setting of AF left atrial catheter ablation will be associated with alow or acceptable risk of major adverse bleeding risks, and low thromboembolic event rates post RF ablation, in accordance with our previous data, and in contrary to the findings of Lakireddy, et al, in their retrospective study published 2012 in JACC. This could lead to widespread utilization of dabigatran etexilate for centers performing a high number of atrial fibrillation and left atrial flutter ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female sex, age 18-85 years.
* Negative pregnancy test for women of childbearing potential
* Planned pulmonary vein isolation by antral radiofrequency or cryoablation for paroxysmal or persistent atrial fibrillation, non-valvular atrial fibrillation (NVAF), or left atrial flutter following prior left atrial ablation procedures
* CHADS2 score of 0-6 or CHADS2-VASc score 0-9
* Vascular hemostasis within 4-6 hours of sheath pull
* Able to give informed consent

Exclusion Criteria:

* Unable to give informed consent
* Currently participating in another clinical treatment trial
* History of hereditary hemophilias
* Presence of active bleeding
* End stage renal disease, CrCl<15 mL/min
* Prior treatment failure of dabigatran (stroke or systemic thromboembolism while on therapeutic dabigatran)
* Known allergic reaction to dabigatran etexilate
* Intolerance to dabigatran, if medication naïve, or other contra-indications as per the USPI.
* Pregnancy
* History of non-compliance
* Inability to follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Ellis, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dabigatran Etexilate Mesylate
Started | 101
Received Initial Dose of Dabigatran | 100
Completed | 94
Not Completed | 7
Not completed — Adverse Event | 6
Not completed — ablation not done, drug not given | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dabigatran Etexilate Mesylate
Number analyzed (Participants) | 100
Age, Continuous [Median (Standard Deviation); unit: years] | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 72
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Major Bleeding Complications in Patients Administered Dabigatran Following RF Ablation.
Time Frame: Within 4 months following procedure (+/- 4 days)
Measure: Number; unit: number of events
Arm/Group | Dabigatran Etexilate Mesylate
Number analyzed (Participants) | 100
number of events | 1

2. Primary Outcome: Frequency of Major Thrombo-embolic Events in Patients Administered Dabigatran Following RF Ablation.
Time Frame: Within 4 months following procedure (+/- 4 days)
Measure: Number; unit: number of events
Arm/Group | Dabigatran Etexilate Mesylate
Number analyzed (Participants) | 100
number of events | 0

3. Secondary Outcome: Dabigatran Serum Drug Levels in Patients Experiencing a Major Bleeding or Thrombo-embolic Event.
Time Frame: Within 4 months following procedure (+/- 4 days)
Population: This measure was removed from the protocol. No blood draws were done on any participants.
Arm/Group | Dabigatran Etexilate Mesylate
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Minor Bleeding Events
Time Frame: Within 4 months following procedure (+/- 4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate Mesylate
Number analyzed (Participants) | 94
Participants | 3

ADVERSE EVENTS:
Arm/Group | Dabigatran Etexilate Mesylate
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 1/100
Other Adverse Events (participants affected / at risk) | 14/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran Etexilate Mesylate (N=100)
Pericardial Effusion with Tamponade (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran Etexilate Mesylate (N=100)
Upper Gi Symptoms (Gastrointestinal disorders) | 5 (5)
Tarry Stools (Gastrointestinal disorders) | 3 (3)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Migraine with Aura (Nervous system disorders) | 1 (1)
Pericardial Pain/Pericarditis (Cardiac disorders) | 1 (1)
Carotid Stenosis/Carotid Endarterectomy (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes